CLINICAL TRIAL: NCT06005922
Title: Investigation of the Effectiveness of Temporomandibular Joint Mobilization and Exercise on Posture, Endurance and Functionality in Individuals With Chronic Neck Pain
Brief Title: The Effectiveness of Temporomandibular Joint Mobilization and Exercise in Individuals With Chronic Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uskudar University (Other)
Responsible Party: Principal Investigator, Dr. Öğr. Üyesi Ömer Şevgin, Asst. Prof. Dr., Uskudar University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Uskudar63
Record Dates: First submitted 2023-08-16; First posted 2023-08-23 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Temporomandibular Joint Disorders; Temporomandibular Joint Dysfunction Syndrome; Neck Pain; Chronic Pain
Keywords: endurance; functionality; joint range of motion
MeSH Terms: conditions — Temporomandibular Joint Disorders; Temporomandibular Joint Dysfunction Syndrome; Neck Pain; Chronic Pain | interventions — Physical Therapy Modalities

STUDY DESIGN:
Intervention Model Description: temporomandibular joint mobilization and temporomandibular joint exercises
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventional physiotherapy methods (Active Comparator): conventional physiotherapy methods
  Interventions: Other: physiotherapy
- temporomandibular joint (TMJ) group (Experimental): conventional physiotherapy methods and temporomandibular joint mobilization and temporomandibular joint exercises
  Interventions: Other: physiotherapy; Other: TMJ exercises

INTERVENTIONS:
Other: physiotherapy — ultrasound hotpack electrotherapy joint range of motion exercises isometric neck exercises stretching exercises
Other: TMJ exercises — tongue relaxation position TMJ isometric strengthening exercises Posture exercises Isometric neck extension in neutral position back extension Strengthening the abdominal muscles Supine dorsal stretch pectoral stretch
  Arms: temporomandibular joint (TMJ) group

SUMMARY:
To examine the effects of temporomandibular joint mobilization and exercises added to the conventional physiotherapy program on posture, functionality and muscular endurance in individuals with chronic neck pain.

DETAILED DESCRIPTION:
Our research is a randomized controlled trial. 50 participants will be included in the study, which will be conducted on individuals aged 18-65 years with chronic neck pain. Participants will be divided into 2 groups as experimental and control groups by simple randomization method. All patients will be treated with conventional physiotherapy methods for 4 weeks and 5 days a week. In addition to conventional treatment, temporomandibular joint mobilization techniques were applied to the experimental group; exercises will be given. In the study, temporomandibular dysfunction (TMD) Pain Screener, Neck Disability Index, and Visual Analog Scale questionnaires will be applied to the patients twice, before and after the treatment. Before and after the treatment, the cervical region's range of motion and muscular endurance will be measured by the physiotherapist. Pre- and post-intervention data were statistically analyzed and compared.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-65,
* Having neck pain lasting longer than 3 months,
* Absence of known systemic disease or trauma history,
* Volunteering to participate in the research.

Exclusion Criteria:

* Having a history of trauma in the areas that are the subject of the study, such as head and neck surgery, upper extremity, thoracic and cervical vertebrae,
* Disc displacement, osteoarthrosis, osteoarthritis signs and symptoms
* Having a neurological-psychiatric diagnosis that may affect the measurement results.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2023-10-20 (Actual); Study Completion 2023-12-03 (Actual)

PRIMARY OUTCOMES:
Neck Disability Index | 6 weeks
  The survey consists of 10 questions. Each question has 5 options. For each question, points are given as A:0, B:1, C:2 D:3 E:4, F:4. 0-4 points are defined as no disability, 5-14 points as mild disability, 15-24 points as moderate disability, 25-34 points as severe disability, 35 or above points as complete disability.

CONTACTS AND LOCATIONS:
Overall Officials: Şeyma DELCEOĞLU, Study Chair — Uskudar University
Locations (1):
- Medicana Hospital, Umraniye, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Calixtre LB, Oliveira AB, de Sena Rosa LR, Armijo-Olivo S, Visscher CM, Alburquerque-Sendin F. Effectiveness of mobilisation of the upper cervical region and craniocervical flexor training on orofacial pain, mandibular function and headache in women with TMD. A randomised, controlled trial. J Oral Rehabil. 2019 Feb;46(2):109-119. doi: 10.1111/joor.12733. Epub 2018 Oct 26. PMID 30307636
- [Background] McCarty WL Jr, Darnell MW. Rehabilitation of the temporomandibular joint through the application of motion. Cranio. 1993 Oct;11(4):298-307. doi: 10.1080/08869634.1993.11677982. PMID 8118901
- [Background] Bernal-Utrera C, Gonzalez-Gerez JJ, Anarte-Lazo E, Rodriguez-Blanco C. Manual therapy versus therapeutic exercise in non-specific chronic neck pain: a randomized controlled trial. Trials. 2020 Jul 28;21(1):682. doi: 10.1186/s13063-020-04610-w. PMID 32723399
- [Background] Reynolds B, Puentedura EJ, Kolber MJ, Cleland JA. Effectiveness of Cervical Spine High-Velocity, Low-Amplitude Thrust Added to Behavioral Education, Soft Tissue Mobilization, and Exercise for People With Temporomandibular Disorder With Myalgia: A Randomized Clinical Trial. J Orthop Sports Phys Ther. 2020 Aug;50(8):455-465. doi: 10.2519/jospt.2020.9175. Epub 2020 Jan 6. PMID 31905097
- [Background] Hidalgo B, Hall T, Bossert J, Dugeny A, Cagnie B, Pitance L. The efficacy of manual therapy and exercise for treating non-specific neck pain: A systematic review. J Back Musculoskelet Rehabil. 2017 Nov 6;30(6):1149-1169. doi: 10.3233/BMR-169615. PMID 28826164